CLINICAL TRIAL: NCT05454033
Title: Multicenter, Evaluator-blind, Randomized, No-treatment Controlled Study to Evaluate the Safety and Effectiveness of JUVÉDERM® VOLITE™ for Correction of Perioral Lines in Chinese Population
Brief Title: A Study to Assess Adverse Events and Effectiveness of Intradermally Injected JUVÉDERM® VOLITE™ Gel Filler in Adult Participants in China With Fine Lines Around the Mouth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M21-528
Record Dates: First submitted 2022-07-08; First posted 2022-07-12 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Perioral Lines
Keywords: Dermal; Dermatology; Aesthetics; Skin Care; Juvederm; Volite; Perioral; Fine Lines; Wrinkles; Frown Lines; Laugh Lines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JUVÉDERM® VOLITE™ (Experimental): Participants in the treatment group will receive a single dose at the study initiation. Participants are eligible for touch up treatment.
  Interventions: Device: JUVÉDERM® VOLITE™
- Control - No Treatment (Other): Participants in the control group will receive no treatment. At Month 2, these participants will have the option to receive the treatment.
  Interventions: Device: JUVÉDERM® VOLITE™; Other: Control

INTERVENTIONS:
Device: JUVÉDERM® VOLITE™ — Injection, intradermal
  Other Names: AGN-8015
Other: Control — No-treatment control
  Arms: Control - No Treatment

SUMMARY:
Facial fine lines and wrinkles are caused by skin thinning, loss of moisture, and loss of elasticity due to factors such as age, ultraviolet (UV) radiation, and environmental exposures. Today, many injectable fillers are used to treat facial aging and correct skin defects. In this study, adverse effects and effectiveness of JUVÉDERM® VOLITE™ will be assessed in correcting perioral lines (around the mouth).

VOLITE is an investigational device being developed for the correction of perioral lines. In this study, participants are placed in 1 of 2 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 3 chance that participants will be assigned to the no-treatment control group. Adult participants seeking improvement of lines, hydration, and skin smoothness in perioral area will be enrolled. Around 198 participants will be enrolled in the study at approximately 12 sites in China.

Participants in the treatment group will receive the initial injection of VOLITE; the control group will receive no treatment, but will have the opportunity to receive VOLITE after 2 months. Participants will be followed up for 12 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend monthly visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Has moderate or severe perioral lines (Perioral Lines at Rest Severity Scale [POLSS] Grades 2 or 3) as assessed by the Evaluating Investigator (EI).
* Participants seeking improvement of lines, hydration, and skin smoothness in perioral area.
* Is able to achieve a 1-point improvement in POLSS score in the judgment of Treating Investigator (TI).
* Participant must be in good health as determined by medical history, vital signs, and TI's judgment, including no known active pandemic infection.

Exclusion Criteria:

* Has a history of anaphylaxis, atopy, or allergy to lidocaine, hyaluronic acid (HA) products, or Streptococcal protein, or is planning to undergo desensitization therapy during the study.
* Has current cutaneous inflammatory or infectious processes (e.g., acne, herpes), abscess, an unhealed wound, angioneurotic edema, cheilitis, or a cancerous or precancerous lesion in the perioral area that could interfere with effectiveness assessments.
* Has a tendency to develop hypertrophic scarring.
* Has impaired cardiac conduction, severely impaired hepatic function, or severe renal dysfunction.
* Has a history of anaphylactic shock.
* Have a history of or currently suffer from autoimmune disease (e.g., rheumatoid arthritis, Crohn's disease) other than Hashimoto's thyroiditis.
* Has porphyria.
* Has a history of skin cancer.
* Has ever received permanent facial implants (e.g., polymethylmethacrylate, silicone, polytetrafluoroethylene) below the subnasale.
* Has ever undergone fat injections or calcium hydroxyapatite below the subnasale.
* Has undergone volume augmentation with semi-permanent soft tissue fillers (e.g., poly-L-lactic acid) within 24 months or temporary soft tissue fillers within 12 months below the subnasale.
* Has undergone treatment with botulinum toxins below the subnasale within 6 months of study entry or is planning to undergo such treatment during the study.
* Has received cosmetic resurfacing below the subnasale within 6 months before enrollment (examples include laser, radiofrequency, dermabrasion, moderate or greater depth chemical peel, or other ablative procedures) or is planning to undergo such treatment during the study.
* Has received mesotherapy or cosmetic treatments below the subnasale within 3 months before enrollment (e.g., photomodulation, intense pulsed light) or is planning to undergo such treatment during the study.
* Has undergone oral surgery (e.g., tooth extraction, aesthetic restoration of front teeth, or implantation in anterior region) within 30 days before enrollment or is planning to undergo any of these procedures during the study.
* Is undergoing orthodontia before enrollment or is planning to undergo it during the study.
* Has changes in use of over-the-counter or prescription oral anti-wrinkle products or topical products below the subnasale within 30 days before enrollment (participants are not eligible for this study if they have begun using any new over-the-counter or prescription oral or topical, anti-wrinkle products below the subnasale within 30 days before enrollment. Participants who have been on a regimen of such products for at least 30 days are eligible for the study if they intend to continue their regimen throughout the study).
* Is on a regimen of anti-coagulation therapy (e.g., warfarin, clopidogrel).
* Is on an ongoing regimen of medications (e.g., aspirin, ibuprofen) or other substances (e.g., herbal supplements with garlic, gingko biloba, or ginseng) known to increase coagulation time within 10 days of undergoing study device injection (study device injection may be delayed as necessary to accommodate this 10-day washout period).
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study.
* Has tattoos, piercings, or scars that would interfere with visual assessment of the perioral lines.
* At TI's discretion, based on participant's safety and/or study integrity, the participant has a condition or is in a situation that, in the TI's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study, such as clinically significant abnormal lab testing results as judged by TI.
* Directly or indirectly involved in the conduct and administration of this study as an investigator, subinvestigator, study coordinator, or other study staff member; employee of the sponsor; first-degree family member, significant other, or relative residing with one of the above persons involved directly or indirectly in the study; or enrolled in the study at another clinical site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
The percentage of participants who achieved at least 1-point improvement from baseline on the Perioral Lines Severity Scale (POLSS) | Up to Month 2
  Responder status based on the Evaluating Investigator's (EI's) live assessment of perioral lines. The POLSS is a 4-point scale from 0 = None, 1 = Mild, 2 = Moderate, to 3 = Severe. An improvement of 1 or more points is an improvement in visibility of perioral lines.

SECONDARY OUTCOMES:
The percentage of participants assessed as "improved" or "much improved" on the Global Aesthetic Improvement Scale (GAIS) by the EI | Up to Month 2
  The Evaluating Investigator (EI) will assess global aesthetic improvement of the perioral area by comparing to frontal and oblique view photographs taken at baseline. The GAIS is a 5-point scale from 2 = Much Improved, 1 = Improved, 0 = No Change, -1 = Worse, to -2 = Much Worse.
The percentage of participants assessed as "improved" or "much improved" on the Global Aesthetic Improvement Scale (GAIS) by the participant | Up to Month 2
  The participant will utilize GAIS to assess global aesthetic improvement of the perioral area by comparing to frontal and oblique view photographs taken at baseline.
The change from baseline on the FACE-Q Appraisal of Lines: Lips questionnaire | Up to Month 2
  The FACE-Q Appraisal of Lines: Lips is a validated scale used to assess the impact of treatment from the participant's perspective. Participants respond to each item on a scale from 1 = Not at all, 2 = A little, 3 = Moderately, to 4 = Extremely.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (11):
- China (11):
  - China-Japan Friendship Hospital /ID# 252139, Beijing, Beijing Municipality
  - Plastic Surgery Hospital(Institute), Cams, Pumc /ID# 231394, Beijing, Beijing Municipality
  - Beijing Hospital /ID# 231393, Beijing, Beijing Municipality
  - Peking University First Hospital /ID# 231392, Xicheng District, Beijing Municipality
  - The Third Affiliated Hospital, Sun Yat-Sen University /ID# 231398, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 231396, Wuhan, Hubei
  - Nanjing Drum Tower Hospital /ID# 231937, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University /ID# 244045, Nanjing, Jiangsu
  - Huashan Hospital, Fudan University /ID# 231395, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University /ID# 231740, Chengdu, Sichuan
  - Hangzhou First People's Hospital /ID# 244111, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M21-528#additional-resources-section